CLINICAL TRIAL: NCT02519790
Title: Optimizing Medication Management for Mothers With Depression
Acronym: OPTI-MOM
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Pittsburgh (Other); The University of Texas Medical Branch, Galveston (Other); Marshfield Clinic (Unknown)
Responsible Party: Principal Investigator, Katherine Wisner, Professor, Northwestern University
Other Study IDs: 1U54HD085601-01 (NIH)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Depression; Pregnancy
Keywords: Pregnancy; Depression; Anxiety; Mental Health; Women
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore the way the antidepressant concentration (amount of medication) in the blood changes due to the physiological changes in the body (i.e., changes in metabolism, hormones and body fluid) during pregnancy and postpartum and the impact of genetic factors on the degree of these changes. Changes in antidepressant concentration are important to monitor, as decreases in antidepressant concentration may lead to less than therapeutic drug levels, which may cause an increase in mood symptoms or recurrence of depressive episodes. Increases in antidepressant concentration have the potential to lead to increased side effects. The study team is hoping to better understand the course of these changes across pregnancy and postpartum and how an individual's genetic makeup impacts these changes with the goal of developing guidelines to optimize antidepressant treatment of pregnant women.

DETAILED DESCRIPTION:
The overarching goal of this The Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) funded U54 Obstetric-Fetal Pharmacology Research Center study is to develop evidence to construct guidelines for the optimal use of selective serotonin reuptake inhibitor (SSRI) antidepressants in pregnant women. The progressive changes in plasma SSRI and metabolite concentrations across pregnancy and after birth will be determined in an observational study. Serial evaluations of depressive and anxiety symptoms and side effects will be obtained to evaluate their association with plasma concentrations at monthly intervals during pregnancy and twice post-birth. To assess the subjects' metabolic phenotypes, subjects have the option to receive a probe drug cocktail, which will be given to evaluate the activities of enzymes involved in antidepressant metabolism during the third trimester (when activity change is maximal) compared to the non-pregnant state after birth.

Additionally, the study team will investigate the impact of genomic variability on inter-individual differences in SSRI dosing, plasma concentrations and pharmacodynamics during pregnancy, with a focus on genes involved in the metabolism and elimination of SSRIs, drug transporters responsible for SSRI access to the central nervous system, and genes encoding critical SSRI targets involved in therapeutic efficacy.

Finally, the study team will determine the maternal-fetal plasma concentrations and pharmacogenetic characteristics associated with neonatal SSRI abstinence syndrome. Maternal and fetal genotypes will be assessed for their relationship to SSRI drug concentrations and neonatal abstinence syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Pregnant, less than or at 18 weeks gestation
* English-speaking
* DSM-IV diagnosis of Major Depressive Disorder (MDD), any subtype
* Medically healthy
* Singleton gestation
* Taking sertraline (Zoloft), fluoxetine (Prozac), or citalopram (Celexa)/escitalopram (Lexapro) and have made the decision to continue this medication throughout pregnancy

Exclusion Criteria:

* DSM-IV diagnosis of bipolar disorder or any psychotic episode
* Substance abuse or dependence in the last 6 months and/or positive urine drug screen
* Primary anxiety disorder without MDD
* EPDS score ≥15, or item 10, self-harm thoughts, is scored 3 "yes, quite often"
* Current use of other therapies for depression, including herbals (such as St. John's Wort)
* Chronic use of drugs for medical disorders except aspirin
* Allergy or adverse reaction to dextromethorphan, omeprazole, midazolam or tolbutamide (exclusion for probe study only; these individuals may still participate in the main study)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample of women taking sertraline (Zoloft), fluoxetine (Prozac), citalopram (Celexa), or escitalopram (Lexapro) in pregnancy and postpartum in areas surrounding Chicago, IL; Pittsburgh, PA and Galveston, TX.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Concentration-to-dose ratio of SSRI in plasma | Every 4 weeks in pregnancy, at delivery, and at 6 and 14 weeks postpartum

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) Scores | Every 4 weeks in pregnancy, at delivery, and at 6 and 14 weeks postpartum
Asberg Side Effects Scale | Every 4 weeks in pregnancy and at 6 and 14 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Wisner, M.D., M.S., Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Marshfield Clinic, Marshfield, Wisconsin